CLINICAL TRIAL: NCT02138955
Title: : A PHASE Ib DOSE ESCALATION STUDY ON THE SAFETY, TOLERABILITY AND ACTIVITY OF LIPOSOMAL CURCUMIN IN PATIENTS WITH LOCALLY ADVANCED OR METASTATIC CANCER
Brief Title: A Phase IB Dose Escalation Study of Lipocurc in Patients With Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SignPath Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lipocurc1002/P-1-010; 0011594-24; SPP1002 (Other: SignPath Pharma,Inc); 2013-001594-24 (EudraCT Number)
Record Dates: First submitted 2014-05-14; First posted 2014-05-15 (Estimated); Last update posted 2022-05-11 (Actual); Status verified 2017-05

CONDITIONS: Patients w/Advanced Cancer That Failed Std of Care Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Liposomeal curcumin ascending dose phase 1b (Experimental)
  Interventions: Drug: Liposomeal curcumin

INTERVENTIONS:
Drug: Liposomeal curcumin

SUMMARY:
This is a single center in patient/outpatient, uncontrolled dose escalating study in cancer patients to evaluate the safety, tolerability and pharmacokinetic (PK) profiles of body surface area adjusted doses of liposomal curcumin administered intravenously as an 8 hour infusion once weekly for 8 weeks.

DETAILED DESCRIPTION:
Patients with solid tumors who either failed to initially respond to approved chemotherapy or who have progressive solid tumor cancers following initial response to approved chemotherapy, are eligible for treatment in this phase 1b trial of ascending doses of intravenous liposomal curcumin following a four week period without previous chemotherapy.The escalating dose range of liposomal curcumin will be from 100mg/M2 to 300 mg/M2 in cohorts of three to 6 patients, and administered over eight hours by a syringe pump weekly for eight weeks. Safety and tolerability will be determined by drug related adverse symptoms(if any), hematologic and serologic signs at each clinic visit and by electronic communication between visits. Pharmacokinetic profiles following infusion of drug will be compared with any adverse changes, and any beneficial subjective or objective responses. When the maximum tolerated dose level is reached in any cohort , another three patients will be accrued at a preceding dose level to assure tolerability in subsequent phase 2 clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients >18 years with a histologically/cytologically confirmed diagnosis of locally advanced or metastatic cancer ,for whom no anti-tumor therapy of proven benefit is available at study enrollment.
* ECOG 0-2.
* Life expectancy of at least 3 months.
* Measurable or non-measurable disease according to RECIST v1.1 criteria.
* Patients should have at least one measurable lesion or disease which is non-measurable but can be clearly be evaluated for response.
* Adequate bone marrow function as evidenced by an absolute neutrophil count :1500 cell/ul.
* Hb greater than 9.5 g/dL and a platelet count greater than 100,000/ uL.
* Renal function >50ml/min with estimated creatinine clearance (eCcr) using the Cockcroft-Gault formula or serum creatinine<1.5 mg/dL.
* Adequate hepatic function as evidenced by serum total bilirubin <3.0 mg/dL, and AST and ALT less than 5 times the upper limit of normal(ULN).
* Signed informed consent.

Exclusion Criteria:

* Patients with lymphoma, hematological cancer or glioblastoma multiforme.
* Active infection, or a fever >38.5C within three days prior to the first day of study drug dosing.
* Current or past history evidence of disease (hemolytic diathesis, hemochromatosis) that could be exacerbated by administering liposomal curcumin.
* Currently on coumadin or coumadin derivatives(oral anticoagulants), or any medications classified as cytochrome p450 inhibitors or inducers.
* Last systemic therapy less than three(3) weeks before (six weeks if treatment was with BCNU or CCNU).
* Unresolved toxicities from prior systemic anti-cancer therapy except symptomatic motor or sensory neuro-toxicities NCI-CTC Grade <2.
* Clinically significant ECG aberrations according to the discretion of the investigator.
* Left ventricular ejection fraction (LVEF) <50%.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03; Primary Completion 2017-11-30 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity with focus on hemolysis | Eight(8) weeks
  The primary objectives of this study are to determine in cancer patients the safety profile of increasing doses of intravenous liposomal curcumin until the maximum tolerated dose (MTD) is determined. This will be done by assessing clinical chemistry, hematology, EKGs and urine analyses, signs and physical symptoms of adverse events.
Determine the maximum tolerated dose of lipocurc | in the cohort after eight ( 8) weeks of treatment
  The primary objectives of this study are to determine in cancer patients the safety profile of increasing doses of intravenous liposomal curcumin until the maximum tolerated dose (MTD) is determined. This will be done by assessing clinical chemistry, hematology, EKGs and urine analyses, signs and physical symptoms of adverse events.
Maximum tolerated dose | eight(8) weeks
  The primary objectives of this study are to determine in cancer patients the safety profile of increasing doses of intravenous liposomal curcumin until the maximum tolerated dose (MTD) is determined. This will be done by assessing clinical chemistry, hematology, EKGs and urine analyses, signs and physical symptoms of adverse events.
Maximum tolerated dose defined by < Grade 1 hematologic toxicity, | Outcome measured weekly x 8 weeks
  The MTD is reached when two or more patients (out of 6) at a dose level experience DLT.

SECONDARY OUTCOMES:
Response by Recist criteria | Eight(8) weeks
  The secondary objectives are to determine the PK profiles of increasing doses, up to the MTD of liposomal curcumin, and to record any evidence of beneficial effect associated with the treatment.
Tumor response by resist criteria | 8 weeks
  The secondary objectives are to determine the PK profiles of increasing doses, up to the MTD of liposomal curcumin, and to record any evidence of beneficial effect associated with the treatment.
Tumor response | Eight weeks
  The secondary objectives are to determine the PK profiles of increasing doses, up to the MTD of liposomal curcumin, and to record any evidence of beneficial effect associated with the treatment.
Benefit | Eight(8) weeks
  The secondary objectives are to determine the PK profiles of increasing doses, up to the MTD of liposomal curcumin, and to record any evidence of related beneficial effect associated with the treatment.
Objective change in measurable tumor size by Resist criteria | once after 8 weeky treatments

OTHER OUTCOMES:
Serologic changes in hepatic, renal, cardiac parameters | weekly x 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard Greil, MD, Principal Investigator — Medicizinische Universitatsklinik Hematologie,Internistische Onkologie
Locations (2):
- Austria (2):
  - 3 Medicizinische Universitatsklinik Hematologie,Internistische Onkologie, Salzburg
  - 3. Medizinische Universitatesclinik, Haematologie, Internistische Onkologie, Salzburg